CLINICAL TRIAL: NCT02757651
Title: Phase I 'Run in' Study Followed by Randomised Phase II Trial Testing Intra-tumoural Hydrogen Peroxide as a Radiation Sensitizer in Women With Locally Advanced/Recurrent Breast Cancer in Terms of Toxicity and Tumour Response
Brief Title: KORTUC: Intra-tumoural Hydrogen Peroxide as a Radiation Sensitizer in Patients With Locally Advanced/Recurrent Breast Cancer in Terms of Toxicity and Tumour Response
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Kortuc, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4502
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Hydrogen Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy + radiation sensitizer (Experimental): Patients in phase I and patients randomised to the test group in phase II will receive standard radiotherapy for breast cancer + a radiation sensitizer
  Interventions: Drug: Hydrogen Peroxide
- Radiotherapy alone (No Intervention): Patients randomised to the control group in phase II will receive standard radiotherapy for breast cancer alone.

INTERVENTIONS:
Drug: Hydrogen Peroxide — Hydrogen Peroxide
  Arms: Radiotherapy + radiation sensitizer

SUMMARY:
This is a study aimed at testing a commonly available and inexpensive chemical (hydrogen peroxide) for safety and activity in sensitising large cancerous lumps in the breast to a standard course of radiotherapy in women with poorly controlled symptoms. Laboratory research and initial clinical trials in Japan suggest that 4 to 6 injections of a radiation sensitiser ('KORTUC') based on very dilute (0.5%) hydrogen peroxide injected into cancers under local anaesthetic twice a week during radiotherapy greatly increases the effectiveness of standard doses of radiotherapy alone. The side effects are limited to mild/moderate discomfort at the injection site for up to 24 hours reported by Japanese breast cancer patients in whom this treatment has been tested. Complete tumour shrinkage in 70/71 (98%) primary breast cancers up to 5 cm diameter have been reported by Japanese collaborators.

DETAILED DESCRIPTION:
PLEASE NOTE: Phase II of this protocol will now be conducted under protocol CCR5119/IRAS 264012 (NCT03946202)

Aim: To test a slow release gel containing a commonly available and inexpensive chemical (hydrogen peroxide) for safety and activity in sensitizing large cancerous lumps in the breast or armpit to a standard 3-week course of radiotherapy in women with poorly controlled symptoms.

Background: Laboratory research and initial clinical trials conducted in Japan raises the possibility that a simple and inexpensive treatment based on a very dilute (0.5%) hydrogen peroxide injected into cancers under local anaesthetic greatly increases the effectiveness of standard doses of radiotherapy. The side effects appear to be limited to mild/moderate discomfort at the injection site for up to 24 hours in one-third of patients. Rapid, complete and durable tumour disappearance has been reported in 49/55 bulky breast cancers in Japanese women treated using this approach, a response that is at least 3 times the success rate of radiotherapy alone in our own patients and in a contemporary Japanese control population. The inventor, Prof Ogawa of Kochi University, has approached the investigators to lead the further clinical evaluation and commercial development, starting with the proposed early phase trials testing safety and anti-cancer activity described below.

Design and methods: After numbing the skin with local anaesthetic, a specialist doctor (radiologist) or trained radiographer will use ultrasound to guide the injection of a small volume of dilute (0.5%) hydrogen peroxide solution into the tumour twice a week during 3 weeks of standard radiotherapy. The drug is suspended in a natural gel (1% sodium hyaluronate, licensed for treating stiff knee joints) that ensures its slow release over 48 hours. The injection procedure lasts for 10-15 minutes altogether. Tiny oxygen bubbles are released from the hydrogen peroxide which help the radiologist guide the injection of drug to the proper places under the skin. The investigators want to test this approach, starting with a careful study of side effects in 12 patients (pilot study) followed by a randomised trial in 84 patients to test activity against cancer (Phase II). Patients participating in Phase II will either have standard radiotherapy or the same radiotherapy plus the drug under test. Neither the patient nor the doctor will choose who has which treatment, which is allocated randomly. Review of the Pilot study data by an independent committee of experts will be completed before starting the phase II (efficacy) study.

Patient and public involvement: Independent Cancer Patient Voice, a patient advocate group in the field of cancer, is collaborating with the investigators on the research plan, commenting and advising on the content and clarity of the written proposal. This group plays a prominent role in promoting UK clinical research, being represented on the Trial Management Groups of several national randomised cancer clinical trials.

Dissemination: The results of this study will be presented at scientific meetings and at meetings of the patient advocate group in order to judge if the results for safety and activity are promising enough to justify taking the research further.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Primary locally advanced breast cancer, or locally recurrent breast cancer with/without metastases
* Radical/high dose palliative radiotherapy required for lifetime control of local morbidities
* Patient physically and mentally fit for radical/high dose palliative radiotherapy
* Target tumour accessible for intra-tumoural injection
* At least one tumour diameter ≥30 mm measurable by ultrasound or magnetic resonance imaging
* Patient available for minimum 3 months follow up post-treatment prior to any surgical resection
* Negative pregnancy test within 7 days of starting radiotherapy in women of child bearing potential and an ability/willingness to protect against pregnancy for 3 months post- radiotherapy
* Patient offers written informed consent

Exclusion Criteria:

* Prior radiotherapy to the target area
* Anatomical location &/or extent of disease difficult to access for safe intra-tumoural drug injections, for example by virtue of contiguous major blood vessels and/or brachial plexus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Phase I: Patient reported maximum intra-tumoural pain intensity over duration of treatment | During radiotherapy
Phase II: Tumour response 3 months post-radiotherapy according to RECIST 1.1 criteria | 3 months months post radiotherapy

SECONDARY OUTCOMES:
Phase I: Proportion of patients with severe pain at any time before and up to 24 hours after any of the KORTUC injections. Server Sever pain is defined as scoring a max grade ≥5 above baseline | During radiotherapy and 3 months post radiotherapy
Phase II: Proportion of patients with severe pain at any time before and up to 24 hours after any of the KORTUC injections. Server pain is defined as scoring a max grade ≥5 above baseline Frequency and duration of pain score ≥1 at each time point | During radiotherapy & 3 and 24 months post radiotherapy
Phase I: Tumour response 3 months post- radiotherapy according to RECIST 1.1 criteria | 3 months post radiotherapy
Phase II: Local progression-free survival at 24 months | 24 months post radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Navita Somaiah, Principal Investigator — The Institute of Cancer Research and The Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom